CLINICAL TRIAL: NCT07395297
Title: The Effectiveness Study of OLE Airway Clearance Therapy in ICU Patients With Pulmonary Infections in EIT Evaluation.
Brief Title: Effectiveness of OLE Airway Clearance Therapy in ICU Patients With Pulmonary Infections
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, wang kaifei, Professer, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2023-270-02
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OLE Airway Clearance Therapy for ICU Patients with Pulmonary Infections (Experimental)
  Interventions: Device: Oscillatory Lung Expansion (OLE) Therapy

INTERVENTIONS:
Device: Oscillatory Lung Expansion (OLE) Therapy — The OLE treatment device is used with synchronized nebulization of 10 ml of 0.9% NaCl solution. The continuous positive airway pressure during the exhalation phase is set to 10-20 cmH₂O, with continuous high-frequency oscillation at a rate of 170-230 times per minute. Each treatment session lasts for 10 minutes. The oxygen therapy parameters are set by the clinician and remain unchanged throughout the experiment.

SUMMARY:
This study aims to explore the application of Electrical Impedance Tomography (EIT) in evaluating the effectiveness of OLE (Oscillatory Lung Expansion) airway clearance therapy for ICU patients with pulmonary infections. The goal is to understand the treatment response differences in patients with various causes of atelectasis (lung collapse). The study will include adult patients diagnosed with pulmonary infections and admitted to the ICU. The primary endpoint of the study is the peak cough flow (CPF), which measures the patient's ability to clear secretions from the lungs through coughing.

ELIGIBILITY:
Inclusion Criteria:

1. Clearly diagnosed with pulmonary infection in the ICU, confirmed by microbiological tests (sputum culture, blood culture, etc.) or imaging tests (chest CT, chest X-ray);
2. Age ≥ 18 years;
3. Respiratory support is oxygen therapy (nasal cannula or face mask oxygen therapy);
4. Sputum volume > 30 ml/day;
5. The patient or their legal representative signs the informed consent form.

Exclusion Criteria:

1. Pregnant or breastfeeding women;
2. Presence of respiratory or circulatory failure (requiring mechanical ventilation or vasopressor support to maintain circulation);
3. Untreated tension pneumothorax;
4. Body Mass Index (BMI) exceeding 50 kg/m²;
5. Rib deformities or severe thoracic deformities;
6. Contraindications for the use of EIT (such as implanted automatic cardiac defibrillators, acute chest trauma, subcutaneous implanted pumps, etc.);
7. Early withdrawal from the study or incomplete clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Cough Peak Flow | Day 1

SECONDARY OUTCOMES:
Lung Ultrasound Score | Day 1
Sputum Viscosity | Day 1
Cough Dysfunction Score | Day 1
Heart rate | Day 1
diastolic pressure | Day 1
systolic pressure | Day 1
Tidal Impedance Variation Before Cough (TIV) | Day 1
End-Expiratory Lung Impedance (EELI) | Day 1
Center of Ventilation (COV) | Day 1
Ventilation Heterogeneity Index (GI) | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No